CLINICAL TRIAL: NCT03712683
Title: Prevalence of Subclinical Hypothyroidism in Women With Unexplained Infertility and the Effect of Thyroxin on Pregnancy Rate
Brief Title: Thyroxin in Subclinical Hypothyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Ariana Jawad, Assistant Professor, Hawler Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HawlerMU2
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Sub Clinical Hypothyroidism; Pregnancy Loss
Keywords: Unexplained Infertility, pregnancy rate,hypothyroidism
MeSH Terms: interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sub clinical hypothyroid women (Experimental): Levothyroxine sodium(Euthyrox 50µg and 25 µg MerckSerono) treatment was initiated and the women were followed in a combined clinic of endocrinologist and Gynecologist.
  2.5 µg of Thyroxine daily was prescribed to women with TSH more than 2.5 mIU/L. Women with TSH more than 4mIU/L were given 50 µg daily . When pregnancy was confirmed Thyroxine was continued till 13 weeks gestation .
  Interventions: Drug: Thyroxine

INTERVENTIONS:
Drug: Thyroxine — Thyroxine was prescribed with the diagnosis of SCH and continued when pregnancy was confirmed
  Other Names: Euthyrox

SUMMARY:
Subclinical hypothyroidism(SCH) is the elevated thyroid stimulating hormone (TSH) with normal free Thyroxine levels and it is a mild or compensated form of primary hypothyroidism. It has been suggested that SCH is more prevalent in infertile women (especially in women with ovulatory disorders.Various rates of SCH was reported in infertile women in different populations

DETAILED DESCRIPTION:
Despite well-established recommendations on screening and treatment of overt hypothyroid in infertile women, there is a controversy regard the treatment of SCH in infertile women .

There are few published data on the prevalence of SCH and the outcome of treatment of SCH in infertile women, many were conducted during IVF cycles . Moreover there are inconsistent results in these studies being authors advised to treat SCH before IVF and some other articles find out no any benefit regarding treatment with Thyroxine in SCH

ELIGIBILITY:
Inclusion Criteria:

1. Unexplained infertility
2. TSH more than 2.5 and normal T3,T4 levels
3. Negative for Anti-thyroid antibodies

Exclusion Criteria:

1. current history of overt hypo or hyperthyroidism
2. recurrent pregnancy loss
3. women having franked causes for infertility like tubal blockage, pelvic inflammatory disease, endometriosis , ,uterine factor
4. Ovarian dysfunction or decreased ovarian reserve
5. abnormal seminal fluid analysis or male factor

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy | 2 years
  Pregnancy was confirmed using human chorionic gonadotropin hormone (hCG) estimation from blood

SECONDARY OUTCOMES:
Miscarriage rate | 13 weeks
  viability and growth of embryos were confirmed by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ariana Kh. Jawad, CABOG, Principal Investigator — Hawler Medical University

IPD SHARING:
Plan to Share IPD: No
Data of the research can be applied on request